CLINICAL TRIAL: NCT06134479
Title: Comparison of Sequential CFA vs CFA +rFSH for Elective Fertility Preservation.. The 2-shot Protocol.
Brief Title: Comparison of Sequential CFA vs CFA +rFSH for Elective Fertility Preservation.
Acronym: 2-Shot
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Santiago Dexeus Font (Other)
Collaborators: Organon (Industry)
Responsible Party: Sponsor
Organization: Fundacion Dexeus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSD-SEQ-2023-09; 2023-506162-31 (EudraCT Number)
Record Dates: First submitted 2023-11-02; First posted 2023-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Fertility
MeSH Terms: interventions — follitropin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 150μg CFA at SD 1 following by rFSH 200IU daily from SD 8 (Active Comparator)
  Interventions: Drug: 150μg CFA (Elonva®) at SD 1 following by rFSH (Puregon®) 200IU daily from SD 8 until the day of the trigger
- 150μg CFA at stimulation day (SD) 1 and 100μg CFA at SD 5 (Experimental)
  Interventions: Drug: 150μg CFA (Elonva®) at stimulation day (SD) 1 and 100μg CFA(Elonva®) at SD 5

INTERVENTIONS:
Drug: 150μg CFA (Elonva®) at stimulation day (SD) 1 and 100μg CFA(Elonva®) at SD 5 — On Day 2 or 3 of the menstrual cycle, a first subcutaneous (SC) injection of corifollitropin alfa (CFA) (Elonva®) 150μg will be administered (stimulation day 1) and a second SC injection of corifollitropin alfa (Elonva®) 100 μg will be administrated on SD 5. Endogenous LH suppression will be accomplished by daily 75μg/day of Desogestrel (Cerazet®) per os, at bedtime, starting on stimulation day 1 and continuing up to the day before of trigger. As soon as 3 follicles ≥ 18 mm are observed by ultrasound, 0.2 mg Triptorelin (Decapeptyl®) will be administered the same day to induce final oocyte maturation. About 34-36 hours thereafter oocyte pick-up will be performed.
  Arms: 150μg CFA at stimulation day (SD) 1 and 100μg CFA at SD 5
Drug: 150μg CFA (Elonva®) at SD 1 following by rFSH (Puregon®) 200IU daily from SD 8 until the day of the trigger — On Day 2 or 3 of the menstrual cycle, a single subcutaneous (SC) injection of corifollitropin alfa (Elonva®) 150μg will be administered (SD 1) and from Day 8 of stimulation a daily SC dose of rFSH (Puregon®) 200IU/day up to the day of Triptorelin (Decapeptyl®) 0.2 mg administration. Endogenous LH suppression will be accomplished by daily 75μg/day of Desogestrel (Cerazet®) per os, at bedtime, starting on stimulation day 1 and continuing up to the day before of trigger. As soon as 3 follicles ≥ 18 mm are observed by ultrasound, 0.2 mg Triptorelin (Decapeptyl®) will be administered the same day to induce final oocyte maturation. About 34-36 hours thereafter oocyte pick-up will be performed.
  Arms: 150μg CFA at SD 1 following by rFSH 200IU daily from SD 8

SUMMARY:
This randomized was designed as non-inferiority trial aiming to compare the number of MII oocytes with 2-shot of Corifollitropin alpha (CFA) sequential administration: 150μg at stimulation day (SD) 1 and 100μg at SD 5 and 1-shot of CFA administration 150μg at SD 1 following by rFSH 200IU daily from SD 8 in women undergoing elective fertility preservation in a progestin-primed ovarian stimulation (PPOS) protocol and GnRH-agonist (GnRH-a) triggering.

ELIGIBILITY:
Inclusion Criteria:

* AFC ≤20
* Anti-Mullerian hormone (AMH) ≤3ng/ml (AMH result of up to one year will be valid)
* Between 18 and 40 years old
* BMI >18 and <30 kg/m2
* Body weight > 50 kg for > 36 years
* Able to come to the Center to comply with the procedures of the study: blood tests, appointments and drug dispensation.

Exclusion Criteria:

* Medically indicated fertility preservation
* AFC > 20
* Polycystic ovarian syndrome (PCOS) according to the Rotterdam criteria
* FSH ≥ 20
* History of untreated autoimmune, endocrine or metabolic disorders
* Contraindication for hormonal treatment
* Recent history of severe disease requiring regular treatment (clinically significant concurrent medical condition that could compromise subject safety or interfered with the trial assessment).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 194 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of MII oocytes retrieved | Trough study completion, an average of 10-20 days.
  Number of MII oocytes retrieved

SECONDARY OUTCOMES:
Total number of oocytes retrieved | Trough study completion, an average of 10-20 days.
  Total number of oocytes retrieved
FSH | Up to oocyte pickup, an average of 10-20 days.
  Endocrine profile FSH
LH | Up to oocyte pickup, an average of 10-20 days.
  Endocrine profile LH
PROGESTERONE | Up to oocyte pickup, an average of 10-20 days.
  Endocrine profile PROGESTERONE
Estradiol | Up to oocyte pickup, an average of 10-20 days.
  Endocrine profile Estradiol
OHSS | Until 15 days after day of oocyte pick-up
  Incidence of OHSS
FertiQoL | from stimulation day 1 until the day of oocyte pick-up,10-20 days after the beggining of the stimulation.
  Quality of life questionnaire "FertiQoL"
Length of stimulation | up to 18 days
  Total days of stimulation
Adverse events | up to 20days
  Frequency of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Quiron Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Begueria R, Garcia D, Vassena R, Rodriguez A. Medroxyprogesterone acetate versus ganirelix in oocyte donation: a randomized controlled trial. Hum Reprod. 2019 May 1;34(5):872-880. doi: 10.1093/humrep/dez034. PMID 30927417
- [Background] Benchabane M, Santulli P, Maignien C, Bourdon M, De Ziegler D, Chapron C, Gayet V. [Corifollitropin alfa compared to daily FSH in controlled ovarian stimulation for oocyte donors]. Gynecol Obstet Fertil Senol. 2017 Feb;45(2):83-88. doi: 10.1016/j.gofs.2016.12.022. Epub 2017 Feb 16. French. PMID 28368800
- [Background] Blockeel C, Polyzos NP, Derksen L, De Brucker M, Vloeberghs V, van de Vijver A, De Vos M, Tournaye H. Administration of corifollitropin alfa on Day 2 versus Day 4 of the cycle in a GnRH antagonist protocol: a randomized controlled pilot study. Hum Reprod. 2014 Jul;29(7):1500-7. doi: 10.1093/humrep/deu105. Epub 2014 May 9. PMID 24813196
- [Background] Cozzolino M, Vitagliano A, Cecchino GN, Ambrosini G, Garcia-Velasco JA. Corifollitropin alfa for ovarian stimulation in in vitro fertilization: a systematic review and meta-analysis of randomized controlled trials. Fertil Steril. 2019 Apr;111(4):722-733. doi: 10.1016/j.fertnstert.2018.11.047. PMID 30929731
- [Background] Croxtall JD, McKeage K. Corifollitropin alfa: a review of its use in controlled ovarian stimulation for assisted reproduction. BioDrugs. 2011 Aug 1;25(4):243-54. doi: 10.2165/11206890-000000000-00000. PMID 21815699
- [Background] Devroey P, Boostanfar R, Koper NP, Mannaerts BM, Ijzerman-Boon PC, Fauser BC; ENGAGE Investigators. A double-blind, non-inferiority RCT comparing corifollitropin alfa and recombinant FSH during the first seven days of ovarian stimulation using a GnRH antagonist protocol. Hum Reprod. 2009 Dec;24(12):3063-72. doi: 10.1093/humrep/dep291. Epub 2009 Aug 14. PMID 19684043
- [Background] Devroey P, Polyzos NP, Blockeel C. An OHSS-Free Clinic by segmentation of IVF treatment. Hum Reprod. 2011 Oct;26(10):2593-7. doi: 10.1093/humrep/der251. Epub 2011 Aug 9. PMID 21828116
- [Background] Drakopoulos P, Vuong TNL, Ho NAV, Vaiarelli A, Ho MT, Blockeel C, Camus M, Lam AT, van de Vijver A, Humaidan P, Tournaye H, Polyzos NP. Corifollitropin alfa followed by highly purified HMG versus recombinant FSH in young poor ovarian responders: a multicentre randomized controlled clinical trial. Hum Reprod. 2017 Nov 1;32(11):2225-2233. doi: 10.1093/humrep/dex296. PMID 29040589
- [Background] Fusi FM, Zanga L, Arnoldi M, Melis S, Cappato M, Candeloro I, Di Pasqua A. Corifollitropin alfa for poor responders patients, a prospective randomized study. Reprod Biol Endocrinol. 2020 Jul 9;18(1):67. doi: 10.1186/s12958-020-00628-6. PMID 32646462
- [Background] Giles J, Alama P, Gamiz P, Vidal C, Badia P, Pellicer A, Bosch E. Medroxyprogesterone acetate is a useful alternative to a gonadotropin-releasing hormone antagonist in oocyte donation: a randomized, controlled trial. Fertil Steril. 2021 Aug;116(2):404-412. doi: 10.1016/j.fertnstert.2021.02.036. Epub 2021 Apr 2. PMID 33814126
- [Background] Hwang JL, Chen SU, Chen HJ, Chen HF, Yang YS, Chang CH, Seow KM, Tzeng CR, Lin YH. Feasibility of corifollitropin alfa/GnRH antagonist protocol combined with GnRH agonist triggering and freeze-all strategy in polycystic ovary syndrome patients. J Formos Med Assoc. 2018 Jun;117(6):535-540. doi: 10.1016/j.jfma.2017.05.009. Epub 2017 Aug 19. PMID 28830648
- [Background] La Marca A, Capuzzo M. Use of progestins to inhibit spontaneous ovulation during ovarian stimulation: the beginning of a new era? Reprod Biomed Online. 2019 Aug;39(2):321-331. doi: 10.1016/j.rbmo.2019.03.212. Epub 2019 Mar 29. PMID 31138494
- [Background] La Marca A, D'Ippolito G. Ovarian response markers lead to appropriate and effective use of corifollitropin alpha in assisted reproduction. Reprod Biomed Online. 2014 Feb;28(2):183-90. doi: 10.1016/j.rbmo.2013.10.012. Epub 2013 Oct 25. PMID 24368127
- [Background] Ledger WL, Fauser BC, Devroey P, Zandvliet AS, Mannaerts BM. Corifollitropin alfa doses based on body weight: clinical overview of drug exposure and ovarian response. Reprod Biomed Online. 2011 Aug;23(2):150-9. doi: 10.1016/j.rbmo.2011.04.002. Epub 2011 Apr 15. PMID 21665541
- [Background] Lerman T, Depenbusch M, Schultze-Mosgau A, von Otte S, Scheinhardt M, Koenig I, Kamischke A, Macek M, Schwennicke A, Segerer S, Griesinger G. Ovarian response to 150 microg corifollitropin alfa in a GnRH-antagonist multiple-dose protocol: a prospective cohort study. Reprod Biomed Online. 2017 May;34(5):534-540. doi: 10.1016/j.rbmo.2017.02.012. Epub 2017 Mar 2. PMID 28285952
- [Background] Loutradis D, Vlismas A, Drakakis P. Corifollitropin alfa: a novel long-acting recombinant follicle-stimulating hormone agonist for controlled ovarian stimulation. Womens Health (Lond). 2010 Sep;6(5):655-64. doi: 10.2217/whe.10.56. PMID 20887164
- [Background] Mahmoud Youssef MA, van Wely M, Aboulfoutouh I, El-Khyat W, van der Veen F, Al-Inany H. Is there a place for corifollitropin alfa in IVF/ICSI cycles? A systematic review and meta-analysis. Fertil Steril. 2012 Apr;97(4):876-85. doi: 10.1016/j.fertnstert.2012.01.092. Epub 2012 Jan 23. PMID 22277766
- [Background] Martinez F, Clua E, Garcia S, Coroleu B, Polyzos NP, Barri PN. Does LH suppression by progesterone-primed ovarian stimulation compared with GnRH antagonist affect live birth rate among oocyte recipients? Reprod Biomed Online. 2020 May;40(5):661-667. doi: 10.1016/j.rbmo.2020.01.016. Epub 2020 Jan 25. PMID 32268981
- [Background] Martinez F, Rodriguez-Purata J, Beatriz Rodriguez D, Clua E, Rodriguez I, Coroleu B. Desogestrel versus antagonist injections for LH suppression in oocyte donation cycles: a crossover study. Gynecol Endocrinol. 2019 Oct;35(10):878-883. doi: 10.1080/09513590.2019.1604661. Epub 2019 May 7. PMID 31062995
- [Background] Massin N. New stimulation regimens: endogenous and exogenous progesterone use to block the LH surge during ovarian stimulation for IVF. Hum Reprod Update. 2017 Mar 1;23(2):211-220. doi: 10.1093/humupd/dmw047. PMID 28062551
- [Background] Polyzos NP, Corona R, Van De Vijver A, Blockeel C, Drakopoulos P, Vloeberghs V, De Vos M, Camus M, Humaidan P, Tournaye H. Corifollitropin alfa followed by hpHMG in GnRH agonist protocols. Two prospective feasibility studies in poor ovarian responders. Gynecol Endocrinol. 2015;31(11):885-90. doi: 10.3109/09513590.2015.1065481. Epub 2015 Jul 14. PMID 26172925
- [Background] Polyzos NP, Devos M, Humaidan P, Stoop D, Ortega-Hrepich C, Devroey P, Tournaye H. Corifollitropin alfa followed by rFSH in a GnRH antagonist protocol for poor ovarian responder patients: an observational pilot study. Fertil Steril. 2013 Feb;99(2):422-6. doi: 10.1016/j.fertnstert.2012.09.043. Epub 2012 Oct 16. PMID 23084565
- [Background] Polyzos NP, Tournaye H, Guzman L, Camus M, Nelson SM. Predictors of ovarian response in women treated with corifollitropin alfa for in vitro fertilization/intracytoplasmic sperm injection. Fertil Steril. 2013 Aug;100(2):430-7. doi: 10.1016/j.fertnstert.2013.04.029. Epub 2013 May 10. PMID 23668992
- [Background] Rombauts L, Talmor A. Corifollitropin alfa for female infertility. Expert Opin Biol Ther. 2012 Jan;12(1):107-12. doi: 10.1517/14712598.2012.641530. Epub 2011 Nov 30. PMID 22129170
- [Background] Seyhan A, Ata B. The role of corifollitropin alfa in controlled ovarian stimulation for IVF in combination with GnRH antagonist. Int J Womens Health. 2011;3:243-55. doi: 10.2147/IJWH.S15002. Epub 2011 Aug 8. PMID 21892335
- [Background] Tsakiridis I, Najdecki R, Tatsi P, Timotheou E, Kalinderi K, Michos G, Virgiliou A, Yarali H, Athanasiadis A, Papanikolaou EG. Evaluation of the safety and efficacy of corifollitropin alfa combined with GnRH agonist triggering in oocyte donation cycles. A prospective longitudinal study. JBRA Assist Reprod. 2020 Oct 6;24(4):436-441. doi: 10.5935/1518-0557.20200033. PMID 32489086
- [Background] Vuong NL, Pham DT, Phung HT, Giang HN, Huynh GB, Nguyen TTL, Ho MT. Corifollitropin alfa vs recombinant FSH for controlled ovarian stimulation in women aged 35-42 years with a body weight >/=50 kg: a randomized controlled trial. Hum Reprod Open. 2017 Nov 28;2017(3):hox023. doi: 10.1093/hropen/hox023. eCollection 2017. PMID 30895237
- [Background] Yovich JL, Keane KN, Borude G, Dhaliwal SS, Hinchliffe PM. Finding a place for corifollitropin within the PIVET FSH dosing algorithms. Reprod Biomed Online. 2018 Jan;36(1):47-58. doi: 10.1016/j.rbmo.2017.09.017. Epub 2017 Oct 31. PMID 29129407
- See also: Related Info — https://www.dexeus.com/